CLINICAL TRIAL: NCT01581346
Title: Pilot Study to Establish an Exercise Intervention in Patients With Lung Cancer
Brief Title: Exercise Study in Patients With Lung Cancer
Acronym: POSITIVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: POSITIVE_II
Record Dates: First submitted 2012-04-05; First posted 2012-04-20 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; exercise intervention; quality of life
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- exercise intervention (Experimental): Pts were instructed to train at least 5 times/ week in the inpatient setting. After discharge pts were instructed to train in a home-based setting at least 3 times/week for a period of 8 weeks.
  Interventions: Other: Exercise intervention

INTERVENTIONS:
Other: Exercise intervention — Pts were instructed to train at least 5 times/ week in the inpatient setting. After discharge pts were instructed to train in a home-based setting at least 3 times/week for a period of 8 weeks.

SUMMARY:
In the course of their disease patients with Non small cell lung cancer (NSCLC) often experience impaired psychological and physical functioning resulting in a reduced quality of life (QoL). The aim of the study is to explore the feasibility and the effects of an eight weeks combined muscle strength and endurance training on physical capacity and QoL.

DETAILED DESCRIPTION:
In this open, prospective, single center study 40 patients (pts) with NSCLC undergoing adjuvant or palliative chemo-/ or radiotherapy are enrolled. Physical status is assessed by using the 6 Minute Walk Test (6MWT) for endurance and by using the Handheld Dynamometer (HHDM) for strength (flexion and extension of elbow, hip and knee). Psychological performance is measured by standardized questionnaires (MFI, FACT-L, PHQ - 9). Data are collected at baseline (T0) and after the 8 weeks sports intervention (T1). Pts are instructed to train at least 5 times/ week in the inpatient setting. After discharge pts are instructed to train in a home-based setting at least 3 times/week for a period of 8 weeks. Feasibility is defined as an adherence of two trainings per week during at least 6 weeks (out of 8 weeks of the intervention).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* histological confirmed diagnosis of Non small cell lung cancer (NSCLC)
* current treatment: chemo-and/or radiotherapy
* age > 18y
* Body Mass Index (BMI) > 18
* written informed consent

Exclusion Criteria:

* acute infection
* immobility > 2 days
* severe neurological impairment
* severe cardiac impairment
* severe pulmonal impairment
* severe renal impairment
* acute bleedings
* alcohol-/drug-abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-03; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
- number of patients who are adherent to the exercise intervention | 8 months
  Adherence is defined as: completion of at least two training sessions per week during minimum six weeks out of eight weeks of the intervention.

SECONDARY OUTCOMES:
- effects of the exercise intervention on psychological symptoms (e.g. quality of life) | 8 months
  Quality of life will be measured by the standardized and validated questionnaire FACT-L;
- effects of the exercise intervention on physical symptoms (muscle strength and endurance) | 8 months
  Muscle strength will be measured by hand held dynamometry and endurance by 6 Minute Walk Test

CONTACTS AND LOCATIONS:
Overall Officials: Michael Thomas, MD, Principal Investigator — Heidelberg University
Locations (1):
- Thoracic Oncology Clinic for Thoracic Diseases, Heidelberg, Germany